CLINICAL TRIAL: NCT06678490
Title: PMCF Registry Study Paclitaxel-eluting Balloon Catheter Support C
Brief Title: Support C Post-Market Registry
Status: Active, not recruiting | Type: Observational
Sponsor: OrbusNeich (Industry)
Collaborators: Eucatech AG (Industry); European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Other Study IDs: DVAL-PLAN-063
Record Dates: First submitted 2024-11-06; First posted 2024-11-07 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Coronary Arteriosclerosis
Keywords: Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Arterioscherosis; Cardiovascular Diseases; Drug Coated Balloon; Ischemic Heart Disease
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Drug Eluting SUPPORT C PTCA balloon catheter: The Drug Eluting SUPPORT C PTCA balloon catheter is indicated for use in patients with symptomatic ischaemic coronary heart disease due to discrete de novo lesions or restenosis of the coronary arteries as well as arterial or venous bypasses.

SUMMARY:
To collect post marketing surveillance data on consecutive patients with coronary heart disease intended to be or treated by the drug eluting Support C PTCA balloon catheter when used according to the Instructions for Use. Data will be collected in order to assess the long term safety and performance of the Support C Drug Coated Balloon (DCB) in routine clinical practice.

DETAILED DESCRIPTION:
This multicenter, prospective registry population consists of consecutive patients with coronary heart disease who undergo percutaneous coronary intervention (PCI) and are intended to be or treated by the Support C Drug Coated Balloon (DCB) according to the Instructions for Use as part of routine clinical care. Approximately 278 patients from 8-12 centers in Europe will be entered into the registry. Patients in the registry are followed for three years. The registry is considered finished when all patients have completed the 36-month follow-up.

A follow-up is scheduled at the following timepoints: immediately post-procedure, 30 days, 6 months, 12 months, 24 months, 36 months. Follow-up is obtained by telephone contact with the patient or at a planned hospital visit.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients intended to be, or treated by Support C DCB as per physicians' decision and according to Instructions for Use (IFU) in the setting of routine clinical care are entered into the registry.

Note:

1. In case of major dissection requiring bailout stenting after DCB use the patients will be included in the registry and followed as per study schedule.
2. If major dissection occurred after lesion preparation, but before DCB use and lesion was stented, the patient will not be included in the registry.

Exclusion Criteria:

* Patients are excluded if ANY of the following additional conditions apply:

  * High probability of non-adherence to the follow-up requirements (due to social, psychological or medical reasons)
  * Currently participating in another investigational drug or device study in which a routine angiographic follow-up is planned
  * A life expectancy of <1year
  * Explicit refusal of participation in the registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic ischemic coronary heart disease due to discrete de novo lesions or restenosis of the coronary arteries as well as arterial or venous bypasses can be included in the study. The vessel diameter must be 2.0 - 4.0 mm.
Sampling Method: Non-Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2025-07-09 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Adjudicated, device-oriented, Target Lesion Failure (TLF) | 12 months post procedure
  Adjudicated, device-oriented, Target Lesion Failure (TLF) where TLF is defined as a composite of cardiac death (CD), non-fatal myocardial infarction (MI) not clearly attributable to a non-target vessel (TV-MI), or clinically driven target lesion revascularization (cd-TLR) (by PCI or coronary artery bypass grafting).

SECONDARY OUTCOMES:
Adjudicated Target Lesion Failure (TLF) | through hospital discharge (expected to be within 24 hours), 30 days, 6 months, 24 months, and 36 months
Each of the components of TLF (cardiac death (CD), non-fatal myocardial infarction not clearly attributable to a non-target vessel (TV-MI), and clinically driven target lesion revascularization (cd-TLR) ) | through hospital discharge (expected to be within 24 hours), 30 days, 6 months, 12 months, 24 months, and 36 months
Adjudicated Target Vessel Failure (TVF) a composite of all Cardiovascular Death (CVD), TV-MI, and clinically driven Target Vessel Revascularization (cd-TVR) | through hospital discharge (expected to be within 24 hours), 30 days, 6 months, 12 months, 24 months, and 36 months
Each of the components of TVF (Cardiovascular Death (CVD), TV-MI, and clinically driven Target Vessel Revascularization (cd-TVR) ) | through hospital discharge (expected to be within 24 hours), 30 days, 6 months, 12 months, 24 months, and 36 months
Adjudicated bleeding Type 3-5 per the Bleeding Academic Research Consortium (BARC) definition | through hospital discharge (expected to be within 24 hours), 30 days, 6 months, 12 months, 24 months, and 36 months
Adjudicated stroke | through hospital discharge (expected to be within 24 hours), 30 days, 6 months, 12 months, 24 months, and 36 months
Adjudicated lesion thrombosis | through hospital discharge (expected to be within 24 hours), 30 days, 6 months, 12 months, 24 months, and 36 months
Device success | Index Procedure
  Successful reaching of the target lesion, successful inflation and deflation of the balloon catheter, and a final residual stenosis after DCB treatment of ≤30% by visual assessment in the presence of grade 3 TIMI (Thrombolysis in Myocardial Infarction) flow, by visual estimation.
Procedure success | Index Procedure
  Procedure success: Successful balloon delivery, deployment and retrieval and no peri-procedural death, TV-MI or TVR.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Alfonso, MD, PhD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (12):
- Czechia (2):
  - Krajska nemocnice Liberec, Liberec
  - Motol University Hospital, Prague
- Germany (4):
  - Katholischen Krankenhaus "St. Johann Nepomuk", Erfurt
  - Evangelisches Krankenhaus Hagen-Haspe gGmbH, Hagen
  - MediClin Herzzentrum Lahr, Lahr
  - Martha Maria Nürnberg, Nuremberg
- National Heart Institute (Institut Jantung Negara), Kuala Lumpur, Malaysia
- Spain (5):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No